CLINICAL TRIAL: NCT01141543
Title: Mobilization of Leukemic Cells Using Plerixafor as Part of a Myeloablative Preparative Regimen for Patients With AML Undergoing Allografting: Assessment of Feasibility and Efficacy
Brief Title: Feasibility and Efficiency Study of Leukemic Cell Mobilization With Plerixafor Injection
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Principal Investigator, Dr. Hans Messner, Physician, University Health Network, Toronto
Other Study IDs: 09-0756-C
Record Dates: First submitted 2010-03-18; First posted 2010-06-10 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Acute Myeloid Leukemia
Keywords: Plerixafor injection
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — plerixafor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- cohort 1: Patients in Cohort 1 will be followed with daily Flowcytometric studies to quantify CXCR4 positive cells.The samples will be obtained before the following doses of FLUDARABINE and BUSULFAN. Eighteen hrs (range 18 -20 hrs) after start of the last dose of FUDARABINE andBUSULFAN and before the first dose of TBI a PB sample as well as bone marrow aspirate and biopsy will be obtained to repeat the studies as conducted prior to the first dose of PLERIXAFOR
  Interventions: Drug: Plerixafor (mozobil)
- Cohort 2: Patients in Cohort 2 will receive the second dose of PLERIXAFOR 24 hrs after the first dose. A PB sample for a CBS and Flowcytometry will be drawn prior to the dose. Nine hrs later a further study sample for Flowcytometry will be obtained prior to administration of the second dose of FLUARABINE and BUSULFAN. Flowcytometric studies will be repeated on day 3 and 4. Eighteen hrs (range 18 - 20 hrs) after start of the last dose of FLUDARABINE and BUSULFAN and before the first dose of TBI a PB sample as well as bone marrow aspirate and biopsy will be obtained to repeat the studies as conducted prior to the first dose of PLERIXAFOR.
  Interventions: Drug: Plerixafor (mozobil)
- cohort 3: Cohort 3: Administration of PLERIXAFOR (240mcg/kg sc) before the first, second, and third dose of FLUARABINE and BUSULFAN
  Interventions: Drug: Plerixafor (mozobil)
- Cohort 4: Administration of PLERIXAFOR (240mcg/kg sc) before all four doses of FLUDARABINE and BUSULFAN
  Interventions: Drug: Plerixafor (mozobil)

INTERVENTIONS:
Drug: Plerixafor (mozobil) — Cohort 1: Administration of PLERIXAFOR (240mcg/kg sc) before the first dose of FLUDARABINE and BUSULFAN Cohort 2: Administration of PLERIXAFOR (240mcg/kg sc) before the first and second dose of FLUDARABINE and BUSULFAN.
  Cohort 3: Administration of PLERIXAFOR (240mcg/kg sc) before the first, second, and third dose of FLUARABINE and BUSULFAN Cohort 4: Administration of PLERIXAFOR (240mcg/kg sc) before all four doses of FLUDARABINE and BUSULFAN
  Other Names: Mozobil

SUMMARY:
The study will be conducted as a single center Phase I/II study to evaluate the safety of administering Plerixafor administered as part of a myeloablative preparative regimen (Institutional Protocol:Fludarabine 50mg/m2/da x 4 days, Busulfan 3.2mg/kg/day x 4 days, TBI 400cGy in divided fractions) for stem cell transplant recipients with AML and to determine whether or not residual leukemic stem cells can be mobilized. Three patients will be enrolled into each of 4 sequential cohorts. Patients in the first cohort will receive 1 dose of Plerixafor (240mcg/kg sc) prior to administration of the first dose of Fludarabine and Busulfan. If tolerated it is planned to escalate the number of Plerixafor doses in the subsequent cohorts to 2. 3. and 4 to be administered before the respective 2nd, 3rd, and 4th dose of chemotherapy.

DETAILED DESCRIPTION:
The study will be conducted as a single center Phase I/II study to evaluate the safety of administering PLERIXAFOR as part of a myeloablative preparative regimen (Institutional Protocol: FBT(400) - FLUDARABINE 50mg/m2/d x 4 days, BUSULFAN 3.2mg/kg/day x 4 days, TBI 400cGy in 2 fractions) for stem cell transplant recipients with Acute Myeloid Leukemia (AML) and to determine whether or not residual leukemic stem cells can be mobilized. Three patients will be enrolled into each of 4 sequential cohorts. Patients in the first cohort will receive 1 dose (240mcg/kg SC) of PLERIXAFOR ( MOZOBIL, formerly known as AMD3100) prior to administration of the first dose of FLUDARABINE and BUSULFAN It is planned to escalate the number of PLERIXAFOR doses in the subsequent cohorts to 2. 3. and 4 to be administered before the respective 2nd, 3rd, and 4th doses of chemotherapy. As primary endpoint the study will establish the toxicity of combined administration of PLERIXAFOR and the preparative regimen at each dose level. Secondary endpoints will include quantification of CXCR4 positive cells and candidates for leukemic disease propagating cells before and after administration of PLERIXAFOR. Mobilized cells will be examined for the ability to undergo apoptosis. Clinical parameters including SAE, OS and LFS are part of the evaluation.

The comparison of cell populations in peripheral blood before and after PLERIXAFOR may facilitate a better definition of minimal residual disease in patients deemed morphologically in a complete remission. The assessment after completion of the preparative regimen will provide a measurement of minimal residual disease prior to the transplant. The assessment of residual leukemic cells with respect to apoptosis will define their responsiveness to the administration of FLUDARABINE and BUSULFAN. The obtained information will facilitate development of a new platform to optimize preparation of patients for a transplant. Eg. Insufficient mobilization of leukemic cells may be addressed in future studies by combining mobilization strategies. Similarly, if cells are shown to be apoptosis resistant one may be able to include apoptosis inducing small molecules.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AML in remission.
* Availability of a suitably matched related or unrelated donor
* Age 18-60 years
* Eligibility for a myeloablative transplant using the Institutional protocols R-FBT(400)-CSMF as preparative regimen for related donors and U-FBT(400)-CP(30)CS for unrelated donors.
* Eligible subjects who are illiterate will be offered participation in the study

Exclusion criteria:

* Patients aged 61years or older
* Patients not eligible for the preparative regimens R-FBT(400)-CSMF or U-FBT(400)-CP(30)CS
* Pregnant or lactating females
* Creatinine of .>2x normal
* Bilirubin, AST, ALT > 2x normal
* MUGA of <50%

Ages: 18 Years to 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study will be performed on patients undergoing myeloablative allogeneic stem cell transplants (PBSC or BM) from related or unrelated donors for the treatment of patients with AML in remission.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2010-05; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Adverse events as a measure of safety and tolerability using Plerixafor in conjunction with a myeloablative preparative regimen for a patients with AML undergoing an allogenic stem cell transplantation. | one year
  As primary endpoint the study is to establish whether or not the administration of Plerixafor during administration of a myeloablative preparative regimen for recipients of allografts can be tolerated.we will complete full protocol with a follow up period of 30 days for first patient than futher patients will be enrolled.Number of Participants with Adverse Events as a Measure of Safety and Tolerability will be evaluated in the study.

SECONDARY OUTCOMES:
Quantification of leukemic progenitor cells after administration of Plerixafor as a myeloablative preparative regimen for a patient with AML undergoing a stem cell transplantation. | one year
  Quantification of CXCR4 positive cells before and after administration of the first and subsequent doses of Plerixafor mesure andNumber of Participants with adverse Events as a measure of safety and tolerability.
Quantification of leukemic progenitor cells after administration of Plerixafor as a myeloablative preparative regimen for a patient with AML undergoing a stem cell transplantation. | One Year
  Qutification of hypermethylation status of Mobilized cells and number of paticipants with adverse event as a measure of safety and Tolerability.
Quantification of leukemic progenitor cells after administration of Plerixafor as a myeloablative preparative regimen for a patient with AML undergoing a stem cell transplantation. | one year
  Qutification of candidates for leukemic cell population s using a marker panel by flowcytometry.
Quantification of leukemic progenitor cells after administration of Plerixafor as a myeloablative preparative regimen for a patient with AML undergoing a stem cell transplantation. | one year
  Qutification of leukemic cells with suitable cytogenic or molrecular markerand number of participants with adverse events measure of safety and tolerability.
Number of Participants with Adverse Events as a Measure of Safety and Tolerability will be evaluated in the study. | one year
  Qutification of normal clonogenic hemopoietic progenitors and number of participants with adverse events as a measure of safety and tolerability.
Number of Participants with Adverse Events as a Measure of Safety and Tolerability will be evaluated in the study. | one year
  overall and Leukemia free survival at 1 year and number of Adverse events as a measure of safety and tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Hans Messner, Ph.D, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Michelis FV, Hedley DW, Malhotra S, Chow S, Loach D, Gupta V, Kim DD, Kuruvilla J, Lipton JH, Viswabandya A, Messner HA. Mobilization of Leukemic Cells Using Plerixafor as Part of a Myeloablative Preparative Regimen for Patients with Acute Myelogenous Leukemia Undergoing Allografting: Assessment of Safety and Tolerability. Biol Blood Marrow Transplant. 2019 Jun;25(6):1158-1163. doi: 10.1016/j.bbmt.2019.01.014. Epub 2019 Jan 14. PMID 30654137